CLINICAL TRIAL: NCT02545530
Title: Transdermal Clonidine on Blood Pressure of Chronic Hemodialysis Patients: A Randomized Crossover Clinical Trial
Brief Title: Transdermal Clonidine in Chronic Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Li Zuo, Head of department of nephrology, Peking University People's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KLD2015.0203
Record Dates: First submitted 2015-09-04; First posted 2015-09-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Renal Dialysis
Keywords: renal dialysis; hypertension; clonidine
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- transdermal clonidine+ (Active Comparator): apply one transdermal clonidine(2.5mg) each week for 4 weeks besides regular antihypertensive agents, reduce oral antihypertensive agents' dosage or type if blood pressure decreased.
  Interventions: Drug: transdermal clonidine
- transdermal clonidine- (No Intervention): regular antihypertensive treatment

INTERVENTIONS:
Drug: transdermal clonidine — 2.5mg/patch per week
  Arms: transdermal clonidine+

SUMMARY:
The majority of chronic hemodialysis patients need a combination of several antihypertensive drugs for adequate BP control. The primary objective of this study is to evaluate whether transdermal clonidine can improve blood pressure control or decrease oral antihypertensive agents type or dosage and the secondary objective is to observe incidence of adverse reactions of transdermal clonidine in chronic hemodialysis patients.

DETAILED DESCRIPTION:
It's a randomised crossover clinical trial. Subjects: chronic hemodialysis patients. All subjects will be randomised to 2 groups. Subjects in first group will receive 4 weeks transdermal clonidine plus regular antihypertensive agents treatments first, 2weeks wash-out then and 4 weeks antihypertensive agents without transdermal clonidine. The other group will receive 4 weeks antihypertensive agents without transdermal clonidine first, 2weeks wash-out then and 4 weeks transdermal clonidine plus regular antihypertensive agents treatments. Ambulatory blood pressure, echocardiography, and biochemistry will be detected.

ELIGIBILITY:
Inclusion Criteria:

1. signed informed consent;
2. age: 18years to 80 years old；
3. on hemodialysis for more than or equal to 3 months, not less than 3 times and 12 hours hemodialysis per week；
4. cardiac function grade I or grade II(NYHA)；
5. Using 1 or more than 1 oral antihypertensive drugs, pre-dialysis systolic blood pressure over 140mmHg or dialysis blood pressure over 90mmHg, post-dialysis systolic blood pressure over 130mmHg or diastolic blood pressure over 80mmHg

Exclusion Criteria:

1. acute infection within 1 month；
2. acute myocardial infarction/cardiac function grade IV/stroke within 3months；
3. LVEF lower than 50% by echocardiography；
4. Dry weight is not suitable by BCM evaluation, more than plus or minus 1kg；
5. Inter-dialysis weight gain exceeds 5% of dry weight；
6. Post-dialysis systolic blood pressure lower than 120mmHg and diastolic blood pressure lower than 70mmHg；
7. Begin or stop recombinant human erythropoietin treatment within 2 weeks before inclusion or 10 weeks after inclusion;
8. Adjust recombinant human erythropoietin dosage to more than 2times or less than half original dosage within 2 weeks before inclusion or 10 weeks after inclusion；
9. The treatment regimen will be amended within 10 weeks and it is expected that the treatment amendment may affect blood pressure；
10. Pregnancy or lactation or planning a pregnancy in 10 weeks；
11. Expected to withdraw hemodialysis treatment in 10 weeks；
12. Allergic to clonidine or its accessories；
13. Undergoing other clinical studies, and the research interventions have an impact on blood pressure；
14. Other clinical conditions that may affect the results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
changes of blood pressure and oral antihypertensive agents' dosage and type | 4 weeks
  mmHg of MAP decreased, changes of total antihypertensive agents' DDD and changes of total antihypertensive agents' types

SECONDARY OUTCOMES:
incidence of adverse effects compared with control group | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Li Zuo, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China